CLINICAL TRIAL: NCT01046318
Title: A Long-term Study of OPC-262 in Patients With Type 2 Diabetes
Brief Title: A Study of OPC-262 in Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kyowa Kirin Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 262-09-004; JapicCTI-090952 (Registry Identifier: JAPIC)
Record Dates: First submitted 2010-01-06; First posted 2010-01-11 (Estimated); Last update posted 2014-01-08 (Estimated); Status verified 2014-01

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- OPC-262 5 mg (Experimental): OPC-262 5 mg will be orally administered once daily fro 52 weeks.
  Interventions: Drug: OPC-262

INTERVENTIONS:
Drug: OPC-262 — OPC-262 5 mg will be orally administered once daily fro 52 weeks.

SUMMARY:
The purpose of this clinical study is to evaluate the safety and efficacy of OPC-262 5 mg in patients with type 2 diabetes by repeated administration orally for 52 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Type 2 diabetes patients with HbA1C above 6.5% and below 10% at both of the time of the 1st and the 2nd screening examinations and who have been undergoing diet and exercise therapies only for at least 8 weeks prior to the 1st screening examination
2. Patients who are capable of giving informed consent
3. Patients who are able to take contraceptive measures to avoid pregnancy of the patient or the patient's partner for the entire study period and for 4 weeks after the study (end of the post-observation period)

Exclusion Criteria:

1. Patients with type 1 diabetes mellitus, patients with diabetes mellitus due to other specified drugs, mechanisms or diseases, and patients with gestational diabetes mellitus
2. Patients with a medical history of diabetic coma
3. Patients with poorly-controlled hypertension
4. Patients with heart failure
5. Patients with a complication of active hepatitis or hepatic cirrhosis
6. Patients undergoing treatment of glomerular diseases other than diabetic nephropathy
7. Patients with a history or complication of malignant tumor

Ages: 20 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2009-11; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Changes in HbA1C from baseline to each visit (OC) and Week 52 (LOCF) | each visit (OC) and Week 52 (LOCF)
Clinical laboratory tests | every 4 weeks

SECONDARY OUTCOMES:
Changes in fasting blood glucose (FBG) from baseline to each visit (OC) and Week 52 (LOCF) | each visit (OC) and Week 52 (LOCF)

CONTACTS AND LOCATIONS:
Locations (3):
- Japan (3):
  - Chubu Region
  - Kanto Region
  - Tohoku Region